CLINICAL TRIAL: NCT01401452
Title: Effectiveness of Adalimumab in Moderate to Severe Plaque Psoriasis Patients With Distinct Co-morbidities
Acronym: EPIC
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Raffeiner GmbH (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-770
Record Dates: First submitted 2011-07-01; First posted 2011-07-25 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-05

CONDITIONS: Moderate to Severe Plaque Psoriasis
Keywords: Monoclonals; Moderate to severe plaque psoriasis; Psoriasis Area & Severity Index (PASI); Adalimumab; Biological disease modifying anti-rheumatic drugs (BDMARD); Co-morbidities; Antibodies; Disease Life Quality Index (DLQI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with psoriasis and at least one co-morbid disease: Participants with moderate to severe plaque psoriasis with at least one co-morbid disease and/or symptom such as hypertension, psoriatic arthritis confirmed by a rheumatologist or other appropriate specialist, obesity, diabetes, metabolic syndrome or depression

SUMMARY:
This multicenter, post marketing observational study (PMOS) was designed to evaluate the effectiveness of adalimumab over a period of 9 months as determined by the Psoriasis Area and Severity Index (PASI) in participants with moderate to severe plaque psoriasis with distinct co-morbidities. Secondary objectives of this study were to measure changes in psychological health via the Dermatology Life Quality Index (DLQI); changes in comorbidities with respect to gender; changes in quality of life using the Short Form Health Survey (SF-36); and evaluation of Minimal Clinically Important Differences (MCID).

DETAILED DESCRIPTION:
Male or female participants ages 18 years of age and older for whom the treating physician had recently prescribed adalimumab were included in this study. Adalimumab was prescribed in accordance with the terms of the local marketing authorization with regards to dose, population, and indication. There were 5 planned visits during the study: baseline (Visit 1), 1 month (Visit 2), 3 months (Visit 3), 6 months (Visit 4), and 9 months (Visit 5).

ELIGIBILITY:
Inclusion Criteria:

Participants for whom adalimumab therapy is indicated and has been prescribed according to the product label and who meet the following criteria:

* Participant age ≥ 18 years
* Participants with moderate to severe plaque psoriasis participants who have at last one co-morbid disease and/or symptom such as hypertension, psoriatic arthritis confirmed by a rheumatologist or other appropriate specialist, obesity, diabetes, metabolic syndrome or depression (diagnosed by a medical specialist for psychology, neurology, or psychiatry)
* Adalimumab naïve participants with moderate to severe plaque psoriasis after unsatisfactory response, non tolerability, or contraindication of systemic therapies such as ciclosporin, methotrexate or PUVA ( psoralen + UVA) or after biological disease modifying anti-rheumatic drugs (bDMARDs) failure (e.g.: infliximab, etanercept or ustekinumab)
* Participants of each country must fulfill any local treatment recommendation for use of bDMARD in psoriasis in their respective country. For Austria: participants must fulfill Austrian Treatment Recommendations for use of bDMARD in psoriasis (Chest X-ray and IGRA* interferon gamma release assay or PPD-skin test negative for tuberculosis)
* Participant is willing to give informed consent to anonymous data collection and their forwarding to AbbVie as well as to informed consent if required in different countries.
* Participant must be able and willing to self-administer adalimumab injections or have a qualified person available to administer Humira® syringe or Humira® Pen injections

Exclusion Criteria:

The following participants will not be included in this observational study:

* Participants who meet contraindications as outlined in the latest version of the Humira syringe® Summary of Product Characteristics (SPC) and Humira Pen® SPC
* Participants participating in another study program or clinical trial
* Participants who have been treated with Humira® before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital, Dermatology
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2011-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Psoriasis and at Least One Co-morbid Disease
Started | 246
Visit 1 (Baseline) | 246
Visit 2 (1 Month) | 225
Visit 3 (3 Months) | 217
Visit 4 (6 Months) | 172
Visit 5 (9 Months) | 175
Completed | 174
Not Completed | 72
Not completed — Adverse reaction | 9
Not completed — Lost to Follow-up | 12
Not completed — Lack of Efficacy | 30
Not completed — Participant developed breast cancer | 1
Not completed — Tx stopped due to financial reasons | 1
Not completed — Tx stopped by psychiatrist | 1
Not completed — No more visits within the 36 wk followup | 4
Not completed — Subject did not come to follow up visits | 2
Not completed — Subject didn't return for routine visits | 1
Not completed — Subject moved to another city | 1
Not completed — Subject's wife wants to get pregnant | 1
Not completed — Psoriatic arthritis | 1
Not completed — Participant stopped Tx | 2
Not completed — Discontinuation for personal reasons | 1
Not completed — Treatment failure | 1
Not completed — Unsatisfactory output | 1
Not completed — Subject withdrew because of Tx success | 1
Not completed — Subject chose to discontinue treatment | 1
Not completed — Participant withdrew consent | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Psoriasis and at Least One Co-morbid Disease
Number analyzed (Participants) | 246
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 153
Duration of psoriasis [Mean (Standard Deviation); unit: years] | 18.6 (13.6)
Number of participants with comorbidities [Number; unit: participants] — Population: Males and females were analyzed separately
  participants
    Female: number analyzed (Participants) | 93
    Female | 93
    Male: number analyzed (Participants) | 153
    Male | 152
Most prevalent co-morbidities among participants in the study [Number; unit: participants]
  Psoriatic arthritis | 114
  Hypertension | 79
  Metabolic syndrome | 72
  Obesity | 64
  Diabetes | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Psoriasis Area and Severity Index 75 (PASI 75) Response at Months 1, 3, 6, and 9
Description: The percentage of participants with a ≥ 75% reduction (improvement) in the Psoriasis Area and Severity Index (PASI) score from baseline was calculated. PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from no symptoms (0), slight (1), moderate (2), marked (3) or very marked (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
Time Frame: Baseline, Months 1, 3, 6, and 9
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Psoriasis and at Least One Co-morbid Disease
Number analyzed (Participants) | 208
percentage of participants
  1 month | 31.3
  3 months: number analyzed (Participants) | 193
  3 months | 52.8
  6 months: number analyzed (Participants) | 154
  6 months | 55.8
  9 months: number analyzed (Participants) | 167
  9 months | 57.5

2. Secondary Outcome: Mean Dermatology Life Quality Index (DLQI) Scores
Description: The DLQI questionnaire asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment- related feelings. Participants respond to 10 questions on a scale from 0 (not at all) to 3 (very much); the range of the total score is 0 to 30. A score of 21 to 30 means that psoriasis has an extremely large effect on the participant's life whereas 0-1 means that the disease has no effect at all.
Time Frame: Baseline, Months 1, 3, 6, and 9
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Psoriasis and at Least One Co-morbid Disease
Number analyzed (Participants) | 238
units on a scale
  Baseline | 12.4 (8.0)
  1 month: number analyzed (Participants) | 214
  1 month | 7.2 (7.1)
  3 months: number analyzed (Participants) | 199
  3 months | 5.4 (6.6)
  6 months: number analyzed (Participants) | 158
  6 months | 4.8 (6.0)
  9 months: number analyzed (Participants) | 169
  9 months | 4.3 (5.7)

3. Secondary Outcome: Percentage of Participants Achieving a Psoriasis Area and Severity Index 50 (PASI 50) Response at Months 1, 3, 6, and 9
Description: The percentage of participants with a ≥ 50% reduction (improvement) in the Psoriasis Area and Severity Index (PASI) score from baseline was calculated. PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from no symptoms (0), slight (1), moderate (2), marked (3) or very marked (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
Time Frame: Baseline, Months 1, 3, 6, and 9
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Psoriasis and at Least One Co-morbid Disease
Number analyzed (Participants) | 208
percentage of participants
  1 month | 51.0
  3 months: number analyzed (Participants) | 193
  3 months | 66.8
  6 months: number analyzed (Participants) | 154
  6 months | 66.9
  9 months: number analyzed (Participants) | 167
  9 months | 72.5

4. Secondary Outcome: Percentage of Participants Achieving a Psoriasis Area and Severity Index 90 (PASI 90) Response at Months 1, 3, 6, and 9
Description: The percentage of participants with a ≥ 90% reduction (improvement) in the Psoriasis Area and Severity Index (PASI) score from baseline was calculated. PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from no symptoms (0), slight (1), moderate (2), marked (3) or very marked (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
Time Frame: Baseline, Months 1, 3, 6, and 9
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Psoriasis and at Least One Co-morbid Disease
Number analyzed (Participants) | 208
percentage of participants
  1 month | 11.5
  3 months: number analyzed (Participants) | 193
  3 months | 38.9
  6 months: number analyzed (Participants) | 154
  6 months | 45.5
  9 months: number analyzed (Participants) | 167
  9 months | 43.7

5. Secondary Outcome: Percentage of Participants Achieving a Psoriasis Area and Severity Index 100 (PASI 100) Response at Months 1, 3, 6, and 9
Description: The percentage of participants with a ≥ 100% reduction (improvement) in the Psoriasis Area and Severity Index (PASI) score from baseline was calculated. PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from no symptoms (0), slight (1), moderate (2), marked (3) or very marked (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
Time Frame: Baseline, Months 1, 3, 6, and 9
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Psoriasis and at Least One Co-morbid Disease
Number analyzed (Participants) | 208
percentage of participants
  1 month | 6.3
  3 months: number analyzed (Participants) | 193
  3 months | 22.3
  6 months: number analyzed (Participants) | 154
  6 months | 32.5
  9 months: number analyzed (Participants) | 168
  9 months | 30.4

6. Secondary Outcome: Mean Health Assessment Questionnaire Short Form 36 (SF-36) Physical Component Summary (PCS) Scores at 1, 3, 6, and 9 Months
Description: The Health Assessment Questionnaire Short Form 36 (SF-36) determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the physical component summary score (PCS) of the SF-36. Items 5-8 primarily contribute to the mental component summary score (MCS) of the SF-36. Scores on each item are summed and averaged (range = 0 "worst"-100 "best"). Increases from baseline indicate improvement. Assessments were conducted at baseline, 1 month, 6 months, and 9 months.
Time Frame: Baseline, Months 1, 3, 6, and 9
Population: Participants with available data. Missing values were imputed if single answers were missing for one dimension.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Psoriasis and at Least One Co-morbid Disease
Number analyzed (Participants) | 232
units on a scale
  Baseline | 46.33 (8.97)
  1 month: number analyzed (Participants) | 207
  1 month | 48.19 (8.87)
  3 months: number analyzed (Participants) | 195
  3 months | 49.54 (8.80)
  6 months: number analyzed (Participants) | 159
  6 months | 49.31 (8.82)
  9 months: number analyzed (Participants) | 162
  9 months | 50.48 (8.24)

7. Secondary Outcome: Mean Health Assessment Questionnaire Short Form 36 (SF-36) Mental Component Summary (MCS) Scores at 1, 3, 6, and 9 Months
Description: as for outcome 6
Time Frame: Baseline, Months 1, 3, 6, and 9
Population: Participants with available data. Missing values were imputed if single answers were missing for one dimension.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Psoriasis and at Least One Co-morbid Disease
Number analyzed (Participants) | 234
units on a scale
  Baseline | 41.35 (11.32)
  1 month: number analyzed (Participants) | 208
  1 month | 45.39 (10.43)
  3 months: number analyzed (Participants) | 195
  3 months | 47.01 (10.25)
  6 months: number analyzed (Participants) | 159
  6 months | 47.92 (10.26)
  9 months: number analyzed (Participants) | 162
  9 months | 48.32 (9.89)

8. Secondary Outcome: Percentage of Participants Achieving Minimal Clinically Important Difference (MCID) in Health Assessment Questionnaire Short Form 36 (SF-36) Physical Component Summary (PCS) Scores at 1, 3, 6, and 9 Months
Description: The Health Assessment Questionnaire Short Form 36 (SF-36) determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the physical component summary score (PCS) of the SF-36. Items 5-8 primarily contribute to the mental component summary score (MCS) of the SF-36. Scores on each item are summed and averaged (range = 0 "worst"-100 "best"). Increases from baseline indicate improvement. Assessments were conducted at baseline, 1 month, 6 months, and 9 months. The percentage of participants achieving MCID in the SF-36 PCS was defined as an increase in PCS of at least 3 points from the baseline score.
Time Frame: Baseline, Months 1, 3, 6, and 9
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Psoriasis and at Least One Co-morbid Disease
Number analyzed (Participants) | 201
percentage of participants
  1 month | 38.3
  3 months: number analyzed (Participants) | 187
  3 months | 52.9
  6 months: number analyzed (Participants) | 150
  6 months | 48.0
  9 months: number analyzed (Participants) | 154
  9 months | 55.2

9. Secondary Outcome: Percentage of Participants Achieving Minimal Clinically Important Difference (MCID) in Health Assessment Questionnaire Short Form 36 (SF-36) Mental Component Summary (MCS) Scores at 1, 3, 6, and 9 Months
Description: The Health Assessment Questionnaire Short Form 36 (SF-36) determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the physical component summary score (PCS) of the SF-36. Items 5-8 primarily contribute to the mental component summary score (MCS) of the SF-36. Scores on each item are summed and averaged (range = 0 "worst"-100 "best"). Increases from baseline indicate improvement. Assessments were conducted at baseline, 1 month, 6 months, and 9 months. The percentage of participants achieving MCID in the SF-36 MCS was defined as an increase in MCS of at least 5 points from the baseline score.
Time Frame: Baseline, Months 1, 3, 6, and 9
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Psoriasis and at Least One Co-morbid Disease
Number analyzed (Participants) | 204
percentage of participants
  1 month | 38.2
  3 months: number analyzed (Participants) | 189
  3 months | 49.7
  6 months: number analyzed (Participants) | 152
  6 months | 52.6
  9 months: number analyzed (Participants) | 155
  9 months | 61.9

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were collected from the time that the informed consent was signed until 70 days after the last dose of study drug (up to 46 weeks). Nonserious adverse events were not collected for this study.
Arm/Group | Participants With Psoriasis and at Least One Co-morbid Disease
Serious Adverse Events (participants affected / at risk) | 13/246
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Psoriasis and at Least One Co-morbid Disease (N=246)
Lymphocytosis (Blood and lymphatic system disorders) | 1
Pneumonia mycoplasmal (Infections and infestations) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Puncture site erythema (General disorders) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Vestibular neuronitis (Infections and infestations) | 1
Priapism (Reproductive system and breast disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.